CLINICAL TRIAL: NCT03731806
Title: Extent of Small Bowel Involvement on Capsule Endoscopy in Newly Diagnosed Patients of Celiac Disease
Brief Title: Capsule Endoscopy in Newly Diagnosed Patients of Celiac Disease
Status: Withdrawn | Type: Observational
Why Stopped: funding for capsule could not be secured
Sponsor: Tazeen Rasheed (Other)
Responsible Party: Sponsor-Investigator, Tazeen Rasheed, Assistant professor, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Other Study IDs: CAP-CELIAC
Record Dates: First submitted 2018-10-25; First posted 2018-11-06 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2019-02

CONDITIONS: Celiac Disease
Keywords: celiac disease; capsule endoscopy
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Celiac Disease is an autoimmune disorder that affects approximately 1% of the world's population 1. The diagnosis of CD requires clinical, histopathological and serological factors 2. Since upper gastrointestinal endoscopy allows only visualization of the small bowel up to the second part of duodenum therefore this study was designed to determine involvement of different segments of small bowel using endoscopic scale by Bonatto MW et al 3 in newly diagnosed patients of celiac disease.

DETAILED DESCRIPTION:
This cross sectional observational study will take place in Medical Unit-II Ruth KM Pfau Civil Hospital Karachi, Pakistan. All newly diagnosed patients of celiac disease between the ages of 8 & 60 years and patients who are currently not on gluten free diet will be included.

Patients having intestinal obstruction, strictures, fistulae, dysphagia, pregnant females will be excluded. Patients having cardiac pacemakers or other implanted electromedical devices and those who are unable to swallow the capsule will also be excluded.

All patients meeting inclusion criteria will be included. Informed consent will be taken from ethics committee. Patients will be provided proper brief information of procedure and confidentiality of the patients will be ensured. Patients will be advised to start clear liquid diet for 24 hours before the procedure. They will be advised to drink Movcol powder 10 sachet in 500ml of water within 20 mins, 12 hours before the procedure. They will be kept nil orally for 08 hours before the procedure. Syrup Infacol (simethicone) 15ml diluted in 50 ml of water will be given 30 mins before the procedure. Patients will be asked to swallow the capsule with 200 ml of water. Patients will be allowed to take food 4 after ingestion of capsule. All patients will be provided with capsule retrieval kit from stool. Patients will be explained to pass any stool after ingestion of capsule till it passed in stool or up to 7 days whichever is earlier. Capsule retrieved will be brought back to investigators for data retrieval from capsule. Reporting will be done by person trained to interpret capsule endoscopy. This will include presence of any pathology, its severity, approximate length and segment of small intestine involved and quality of bowel preparation.

Categorical data will be presented as frequency and percentage, e.g., gender, findings of capsule endoscopy like, bowel preparation, mosaic pattern,ulcers, erythema, telangiectasia etc. Quantitative data will be presented as mean with standard deviation, e.g., age. Involvement of different segments of small intestine (duodenum, jejunum and Ileum) will be documented. Categorical data will be compared on gender by Chi-square test and quantitative data will be analyzed by student's t-test. Significance level will be set at ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

1. All newly diagnosed patients of celiac disease between the ages of 8 & 60 years.
2. Patients who are currently not on gluten free diet.

Exclusion Criteria:

1. Patients having intestinal obstruction, strictures, fistulae, dysphagia will be excluded.
2. Pregnant females will be excluded.
3. Patients having cardiac pacemakers or other implanted electromedical devices.
4. Unable to swallow capsule.

Ages: 8 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients of celiac disease presenting to the OPD or admitted in Medical wards of Dr.Ruth KM Pfau ,Civil Hospital Karachi, Pakistan.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Grading of Celiac Disease on Capsule Endoscopy using Bonatto Classification | 8 hours
  Bonatto Endoscopic Classification of Celiac
  * 0 = Normal
  * I = Mostly regular villi, some foci, no mosaic pattern
  * II = Agglutinated but visible villi, mosaic pattern
  * III = Mosaic pattern, absence of villi

CONTACTS AND LOCATIONS:
Overall Officials: Bader F Zuberi, FCPS, Study Chair — Dow University of Health Sciences
Locations (1):
- Ruth KM Pauf Civil Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tennyson CA, Green PH. The role of capsule endoscopy in patients with nonresponsive celiac disease. Gastrointest Endosc. 2011 Dec;74(6):1323-4. doi: 10.1016/j.gie.2011.07.021. No abstract available. PMID 22136777
- [Background] Lujan-Sanchis M, Perez-Cuadrado-Robles E, Garcia-Lledo J, Juanmartinena Fernandez JF, Elli L, Jimenez-Garcia VA, Egea-Valenzuela J, Valle-Munoz J, Carretero-Ribon C, Fernandez-Urien-Sainz I, Lopez-Higueras A, Alonso-Lazaro N, Sanjuan-Acosta M, Sanchez-Ceballos F, Rosa B, Gonzalez-Vazquez S, Branchi F, Ruano-Diaz L, Prieto-de-Frias C, Pons-Beltran V, Borque-Barrera P, Gonzalez-Suarez B, Xavier S, Arguelles-Arias F, Herrerias-Gutierrez JM, Perez-Cuadrado-Martinez E, Sempere-Garcia-Arguelles J. Role of capsule endoscopy in suspected celiac disease: A European multi-centre study. World J Gastroenterol. 2017 Jan 28;23(4):703-711. doi: 10.3748/wjg.v23.i4.703. PMID 28216978
- [Background] Bonatto MW, Kotze L, Orlandoski M, Tsuchyia R, de Carvalho CA, Lima D, Kurachi G, Orso IR, Kotze L. Endoscopic evaluation of celiac disease severity and its correlation with histopathological aspects of the duodenal mucosa. Endosc Int Open. 2016 Jul;4(7):E767-77. doi: 10.1055/s-0042-108190. Epub 2016 Jun 29. PMID 27556094